CLINICAL TRIAL: NCT04013854
Title: Adjuvant Nivolumab or Ipilimumab + Nivolumab Determined By Pathological Response To A Single Dose Of Neoadjvuant Nivolumab
Brief Title: Adjuvant Treatment Determined By Pathological Response To Neoadjvuant Nivolumab
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 02619
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Melanoma Stage III; Melanoma
Keywords: nivolumab; ipilimumab; adjuvant; neoadjuvant; surgery
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A: Adjuvant Nivolumab (Complete Pathological Response) (Active Comparator): 480 mg IV for up to one year
  Interventions: Drug: nivolumab
- Arm B: Adjuvant Nivolumab (Less than Complete Response) (Active Comparator): 480 mg IV for up to one year
  Interventions: Drug: nivolumab
- Arm C: Adjuvant Combination (Less than Complete Response) (Experimental): ipilimumab (1mg/kg) plus nivolumab (3mg/kg) for 4 doses and then nivolumab (480 mg) alone for a total of one year
  Interventions: Drug: nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: nivolumab — All arms will receive a pre-surgery dose of nivolumab (480 mg IV). Post-surgery nivolumab doses will be determined by pathologic response and randomization.
Drug: Ipilimumab — Only subjects who fail to achieve a complete, or near complete, pathological response, and are then randomized to Arm C will receive Ipilimumab (1 mg/kg) )
  Arms: Arm C: Adjuvant Combination (Less than Complete Response)

SUMMARY:
Subjects with resectable melanoma will receive neoadjuvant nivolumab followed by surgical resection. Post-operatively, subjects will receive open-label treatment with up to 1 year of adjuvant nivolumab or ipilimumab plus nivolumab as determined by pathologic response at the time of resection.

DETAILED DESCRIPTION:
Subjects with Stage III resectable melanoma will receive one dose of nivolumab 480 mg IV, then undergo standard definitive surgery approximately 4 weeks after the initial dose of nivolumab. Post-operatively, subjects will receive open-label treatment with up to 1 year of adjuvant nivolumab 480 mg IV every 4 weeks or ipilimumab plus nivolumab, as determined by pathologic response at the time of resection. Subjects with pathologic complete response or near pathologic complete response (PathCR/nearCR) (Arm A) receive adjuvant nivolumab for up to one year. Subjects with <PathCR/nearCR are randomized 1:2 to either adjuvant nivolumab (480 mg) for up to one year (Arm B) or adjuvant ipilimumab (1mg/kg) plus nivolumab (3mg/kg) for 4 doses and then nivolumab (480 mg) alone for a total of one year (Arm C).

ELIGIBILITY:
Inclusion Criteria:

* The subject must have clinical stage III resectable melanoma per investigator. Subjects may not have a diagnosis of uveal or mucosal melanoma.
* Either the subject or the subject's legally authorized representative must be willing and able to provide written informed consent before the performance of any protocol-related procedures.
* The subject must be ≥18 years of age on day of signing informed consent.
* The subject must have a performance status of 0 or 1 on the ECOG Performance Scale.
* The subject must demonstrate adequate organ function as defined in Table 1; all screening labs must be performed within 28 days of treatment initiation.

  * Hematologic System: Absolute neutrophil count (ANC) ≥1500/mcL; Platelets ≥100,000/mcL; Hemoglobin ≥9 g/dL or ≥5.6 mmol/L
  * Renal System: Serum creatinine OR measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR ≥50 mL/min for subject with creatinine levels >1.5 X institutional ULN
  * Hepatic System: Serum total bilirubin ≤1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels >1.5 ULN; AST (SGOT) and ALT (SPGT) ≤2.5 X ULN OR ≤5 X ULN for subjects with liver metastases
* A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies: A.) Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR B.) A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and is willing to use a highly effective method of contraception or abstain from heterosexual intercourse for at least 2 weeks prior to the time of first dose of study medication through 5 months after the last dose of study medication.
* Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication.
* Male subjects must agree to follow the contraceptive guidance in Appendix 3 starting with the first dose of study medication, while on study, through 7 months after the last dose of study medication.

Exclusion Criteria:

* Subject has unresectable disease; i.e. in the opinion of the surgical oncologist, all of the subject's melanoma cannot be completely removed with a clear margin.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137), interferon, high dose IL-2 or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to the first dose of study drug. Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy are an exception to this criterion.
* If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
* Subject has received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including G-CSF, GM-CSF or recombinant erythropoietin) within 4 weeks to the first dose of study drug.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or requires active treatment. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has active autoimmune disease that has required systemic treatment in the past 3 months (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has evidence of active interstitial lung disease or a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Patients known to be positive for Human Immunodeficiency Virus (HIV) if they have a CD4 count of less than 350 mm3 and a serum HIV viral load > 25,000 IU/mL
* Has active Hepatitis B infection or active Hepatitis C virus infection as determined by medical record review.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 5 months, if female, or 7 months, if male, after the last dose of investigational drug.
* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival | 1 year
  Recurrence-free survival (RFS) is defined as the time from date of surgery to date of disease recurrence, death due to any cause or most recent follow-up documenting freedom from recurrence (i.e., scan date).

SECONDARY OUTCOMES:
Frequency and Incidence of Adverse Events | Up to 13 months
  Toxicity will be determined by scoring treatment-related AEs and SAEs. CTCAE version 5.0 grades will be employed.
Pathological Response Rate | Approximately 4 weeks
  The number of subjects with pathologic complete response (CR) or near CR defined by less than 10% viable tumor cells will be determined for subjects who received 1 dose of neoadjuvant Nivolumab and underwent definitive surgery. PathCR/nearCR rate is defined as the percentage of treated subjects who achieve PathCR/nearCR
Overall Survival | Up to 7 Years
  Overall survival (OS) is defined as the time from date of surgery to date of death due to any cause or last subject contact alive.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Duke Cancer Institute, Durham, North Carolina
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Abramson Cancer Center, University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weber J, Mandala M, Del Vecchio M, Gogas HJ, Arance AM, Cowey CL, Dalle S, Schenker M, Chiarion-Sileni V, Marquez-Rodas I, Grob JJ, Butler MO, Middleton MR, Maio M, Atkinson V, Queirolo P, Gonzalez R, Kudchadkar RR, Smylie M, Meyer N, Mortier L, Atkins MB, Long GV, Bhatia S, Lebbe C, Rutkowski P, Yokota K, Yamazaki N, Kim TM, de Pril V, Sabater J, Qureshi A, Larkin J, Ascierto PA; CheckMate 238 Collaborators. Adjuvant Nivolumab versus Ipilimumab in Resected Stage III or IV Melanoma. N Engl J Med. 2017 Nov 9;377(19):1824-1835. doi: 10.1056/NEJMoa1709030. Epub 2017 Sep 10. PMID 28891423
- [Background] Eggermont AMM, Blank CU, Mandala M, Long GV, Atkinson V, Dalle S, Haydon A, Lichinitser M, Khattak A, Carlino MS, Sandhu S, Larkin J, Puig S, Ascierto PA, Rutkowski P, Schadendorf D, Koornstra R, Hernandez-Aya L, Maio M, van den Eertwegh AJM, Grob JJ, Gutzmer R, Jamal R, Lorigan P, Ibrahim N, Marreaud S, van Akkooi ACJ, Suciu S, Robert C. Adjuvant Pembrolizumab versus Placebo in Resected Stage III Melanoma. N Engl J Med. 2018 May 10;378(19):1789-1801. doi: 10.1056/NEJMoa1802357. Epub 2018 Apr 15. PMID 29658430
- [Background] Huang AC, Orlowski RJ, Xu X, Mick R, George SM, Yan PK, Manne S, Kraya AA, Wubbenhorst B, Dorfman L, D'Andrea K, Wenz BM, Liu S, Chilukuri L, Kozlov A, Carberry M, Giles L, Kier MW, Quagliarello F, McGettigan S, Kreider K, Annamalai L, Zhao Q, Mogg R, Xu W, Blumenschein WM, Yearley JH, Linette GP, Amaravadi RK, Schuchter LM, Herati RS, Bengsch B, Nathanson KL, Farwell MD, Karakousis GC, Wherry EJ, Mitchell TC. A single dose of neoadjuvant PD-1 blockade predicts clinical outcomes in resectable melanoma. Nat Med. 2019 Mar;25(3):454-461. doi: 10.1038/s41591-019-0357-y. Epub 2019 Feb 25. PMID 30804515
- [Derived] Gorry C, McCullagh L, O'Donnell H, Barrett S, Schmitz S, Barry M, Curtin K, Beausang E, Barry R, Coyne I. Neoadjuvant treatment for stage III and IV cutaneous melanoma. Cochrane Database Syst Rev. 2023 Jan 17;1(1):CD012974. doi: 10.1002/14651858.CD012974.pub2. PMID 36648215